CLINICAL TRIAL: NCT04388709
Title: A Randomized Phase 2 Trial of Peginterferon Lambda-1a (Lambda) for the Treatment of Hospitalized Patients Infected With SARS-CoV-2 With Non-critical Illness
Brief Title: Interferon Lambda Therapy for COVID-19
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to the number of competing trials at their site, the study team has closed enrollment and withdrawn this trial.
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Eiger BioPharmaceuticals (Industry)
Responsible Party: Principal Investigator, Thomas Marron, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 20-0820
Record Dates: First submitted 2020-05-12; First posted 2020-05-14 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: SARS-CoV-2
Keywords: Peginterferon lambda-1a; Lambda; SARS-CoV-2
MeSH Terms: interventions — peginterferon lambda-1a; Interferon Lambda

STUDY DESIGN:
Intervention Model Description: Cohort A: Peginterferon lambda-1a (Lambda) 180mcg subcutaneous injection once Cohort B: Best supportive care
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Peginterferon lambda-1a (Experimental): Peginterferon lambda-1a (Lambda) 180mcg subcutaneous injection once
  Interventions: Drug: Peginterferon Lambda-1A
- Best supportive care (No Intervention): Best supportive care

INTERVENTIONS:
Drug: Peginterferon Lambda-1A — Peginterferon lambda-1a (Lambda) 180mcg subcutaneous injection once
  Other Names: Lambda; Interferon Lambda
  Arms: Peginterferon lambda-1a

SUMMARY:
The main purpose of this research study is to test the safety and effectiveness of an investigational drug peginterferon lambda-1a in treating COVID-19.

DETAILED DESCRIPTION:
Primary Objective: Determine efficacy of pegylated interferon lambda as measured by clinical improvement. This will be defined as improvement in supplemental oxygen requirement.

Secondary Objectives:

* Determine safety and tolerability of pegylated interferon lambda
* Days with fever
* Time to resolution of fever
* Rate of progression to requiring critical care
* Overall survival
* Time to discharge

Exploratory Objectives: Determining the effect systemically on inflammatory markers in the blood, as well as viral load.

Diagnosis and Main Inclusion Criteria: Patients must have a confirmed diagnosis of infection with SARS-CoV-2 and be receiving supplemental oxygen. Many patients may be receiving hydroxychloroquine with or without other antimicrobials.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of SARS-CoV-2
* Hospitalization due to diagnosis with SARS-CoV-2
* Sp02 < 93% on ambient air or PaO2/FiO2 < 300 mmHg and requires supplemental oxygen

Exclusion Criteria:

* Patients must not be pregnant or nursing
* Patients cannot be admitted to intensive care unit at time of admission or require positive pressure ventilation
* Patients cannot be requiring continuous supplemental oxygen normally (pre-SARS-CoV-2)
* Patient is receiving steroids >1mg/kg
* Has diagnosis of primary immunodeficiency
* Has active autoimmune disease that has required systemic treatment in the past year
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial
* Patients with ferritin >2000ng/mL and/or C-reactive protein >100mg/L
* History of allogeneic hematopoietic cell transplantation or solid organ transplantation
* Childs-Pugh class B or C cirrhosis or class A if portal hypertension is present
* Documented allergic or hypersensitivity response to protein therapeutics
* No serious disease requiring mechanical ventilation at time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-02-05 (Actual); Study Completion 2021-02-05 (Actual)

PRIMARY OUTCOMES:
Number of participants with resolution of hypoxia | 7 days
  The clinical improvement as defined as resolution of hypoxia requiring supplemental oxygen to maintain SpO2>92% at 7 days.

SECONDARY OUTCOMES:
Number of adverse events. | until 90 days after receipt of treatment
  Number of Grade 3 or 4 adverse events as determined by the DAIDS criteria over the course of 3 months from initiation of trial to measure safety and tolerability of pegylated interferon lambda. Information on adverse events will be collected during hospitalization and then as an outpatient until 90 days from the time of receipt of treatment.
Days with fever | during hospitalization, average of 7 days
  Number of days participant has a fever. Information on fever will be collected during hospitalization. Cessation of fever is defined as the beginning of the first 48 hour period without fever without the use of antipyretic drug.
Time to resolution of fever | during hospitalization, average of 7 days
  This is defined as time from initial treatment with investigational agent, to the cessation of fever, defined as the beginning of the first 48 hour period without fever without the use of antipyretic drug.
Rate of progression to requiring critical care | during hospitalization, average of 5 days
  Defined as time from initial treatment with investigational agent to deterioration of clinical condition necessitating transfer to a critical care unit and/or intubation.
Overall survival | until 90 days after receipt of treatment
  Information on survival will be collected during hospitalization and then, for those patients discharged, will be collected as an outpatient until 90 days from the time of receipt of treatment
Time to discharge | average of 7 days
  This is defined as the amount of time (in days or fraction thereof) between the receipt of investigational agent and discharge from The Mount Sinai Hospital to home or nursing home, or censoring at time of death.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Marron, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee JS, Shin EC. The type I interferon response in COVID-19: implications for treatment. Nat Rev Immunol. 2020 Oct;20(10):585-586. doi: 10.1038/s41577-020-00429-3. PMID 32788708